CLINICAL TRIAL: NCT02848131
Title: Senescence, Frailty, and Mesenchymal Stem Cell Functionality in Chronic Kidney Disease: Effect of Senolytic Agents
Brief Title: Senescence in Chronic Kidney Disease
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, LaTonya J. Hickson, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-005843
Record Dates: First submitted 2016-03-22; First posted 2016-07-28 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Observational (No Intervention): Observational Only
- Group 2: Dasatinib & Quercetin (Active Comparator): The drugs dasatinib and quercetin will be used in this arm
  Interventions: Drug: Group 2: Dasatinib; Drug: Group 2: Quercetin

INTERVENTIONS:
Drug: Group 2: Dasatinib — Dasatinib - take one 100 mg tablet by mouth once daily for 3 consecutive days.
  Other Names: Sprycel
  Arms: Group 2: Dasatinib & Quercetin
Drug: Group 2: Quercetin — Quercetin - take four 250 mg capsules daily (total 1000 mg daily) for 3 consecutive days.
  Arms: Group 2: Dasatinib & Quercetin

SUMMARY:
The study goal is to assess the effect of senescent cell clearance on senescence burden, physical ability or frailty, and adipose tissue-derived mesenchymal stem cell (MSC) functionality in patients with chronic kidney disease (CKD).

DETAILED DESCRIPTION:
The proposed studies will examine cellular senescence and the effect of senolytic therapy on senescent cell burden, frailty, and adipose-derived mesenchymal stem cell function in individuals with diabetic chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80 years
2. Chronic kidney disease estimated glomerular filtration rate (eGFR) 15-45 ml/min/1.73m2
3. Diabetes mellitus and taking diabetes medications

Exclusion Criteria:

1. Concomitant glomerulonephritis,
2. Nephrotic syndrome,
3. Solid organ transplantation,
4. Autosomal dominant or recessive polycystic kidney disease,
5. Known renovascular disease,
6. Pregnancy,
7. Active immunosuppression therapy,
8. Hemoglobin A1c≥10% at screening,
9. History of active substance abuse (including alcohol) within the past 2 years,
10. Current alcohol abuse (>3 alcoholic beverages/day or >21 per week),
11. Body weight >150 kg or body mass index>50
12. Human immunodeficiency virus infection
13. Active hepatitis B or C infection
14. Tyrosine kinase inhibitor therapy
15. Known hypersensitivity or allergy to dasatinib or quercetin
16. Inability to give informed consent
17. Uncontrolled systemic lupus erythematosus
18. Uncontrolled pleural/pericardial effusions or ascites
19. New invasive cancer except non-melanoma skin cancers
20. Invasive fungal or viral infection
21. Inability to tolerate oral medications
22. Total bilirubin>2x upper limit of normal
23. Subjects taking medications that are sensitive to substrates or substrates with a narrow therapeutic range for CYP3A4, CYP2C8, CYP2C9, or CYP2D6 or strong inhibitors or inducers of CYP3A4 (e.g. cyclosporine, tacrolimus or sirolimus). If antifungals are absolutely necessary from an infectious disease perspective, then they will be allowed only if the levels are therapeutic.
24. Subjects on strong inhibitors of CYP3A4.
25. Subjects on therapeutic doses of anticoagulants (Warfarin (Coumadin);Rivaroxaban (Xarleto); Apixaban (Eliquis); Dabigatran (Pradaxa, Prazaxa) or Other).
26. Subjects on antiplatelet agents ((Clopidogrel (Plavix); Dipyridamole + Asprin (Aggrenox); Ticagrelor (Brilinta); Prasugrel (Effient); Ticlopidine (Ticlid) or Other) who are unable or unwilling to reduce or hold therapy prior to and during the 3-day drug dosing. Subjects may continue their previous regimen on day 4.
27. Subjects on quinolone antibiotic therapy for treatment or for prevention of infections within 10 days
28. Subjects taking H2-antagonists or proton pump inhibitors and unwilling to discontinue therapy 1 week prior and 2 weeks following enrollment.
29. Corrected QT interval (QTc)>450 msec
30. Presence of any condition that the Investigator believes would put the subject at risk or would preclude the patient from successfully completing all aspects of the trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in proportion of senescent cells (representing the total senescent cell burden) present | Baseline, Day 14
  Assessment of senescence markers in skin, fat, and/or blood at baseline and day 14.

SECONDARY OUTCOMES:
Change in proportion of senescent mesenchymal stem cells present | Baseline, Day 14
  Assessment of senescence markers in mesenchymal stem cells at baseline and day 14.
Change in mesenchymal stem cell function | Baseline, Day 14
  Assessment of functional studies in mesenchymal stem cells at baseline and day 14. Number of subjects with change in stem cell function related to treatment.
Change in Frailty index score | Baseline, Day 14
  Assessment by Fried and other frailty criteria at baseline and day 14.
Change in kidney function | Baseline, Day 14, Month 4, Month 12
  Assessment by estimated and measured glomerular filtration rate at baseline, day 14, month 4, and month 12.

CONTACTS AND LOCATIONS:
Overall Officials: LaTonya J Hickson, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bian X, Snow ZK, Zinn CJ, Gowan CC, Conley SM, Bratulin AL, Elhusseiny KM, Miller J, Tchkonia T, Kirkland JL, Lerman LO, Hickson LJ. Activin A Antagonism with Follistatin Reduces Kidney Fibrosis, Injury, and Cellular Senescence-Associated Inflammation in Murine Diabetic Kidney Disease. Kidney360. 2025 Mar 28;6(8):1278-1291. doi: 10.34067/KID.0000000776. PMID 40152935
- [Derived] Hickson LJ, Langhi Prata LGP, Bobart SA, Evans TK, Giorgadze N, Hashmi SK, Herrmann SM, Jensen MD, Jia Q, Jordan KL, Kellogg TA, Khosla S, Koerber DM, Lagnado AB, Lawson DK, LeBrasseur NK, Lerman LO, McDonald KM, McKenzie TJ, Passos JF, Pignolo RJ, Pirtskhalava T, Saadiq IM, Schaefer KK, Textor SC, Victorelli SG, Volkman TL, Xue A, Wentworth MA, Wissler Gerdes EO, Zhu Y, Tchkonia T, Kirkland JL. Senolytics decrease senescent cells in humans: Preliminary report from a clinical trial of Dasatinib plus Quercetin in individuals with diabetic kidney disease. EBioMedicine. 2019 Sep;47:446-456. doi: 10.1016/j.ebiom.2019.08.069. Epub 2019 Sep 18. PMID 31542391
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT02848131/Prot_SAP_001.pdf